CLINICAL TRIAL: NCT04671966
Title: Mechanism and Modulation of Sex Differences in Myocardial Steatosis Induced Left Ventricular Dysfunction
Brief Title: Sex Differences in Myocardial Steatosis Induced Left Ventricular Dysfunction
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STU 112017-013
Record Dates: First submitted 2020-12-03; First posted 2020-12-17 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Heart Diseases; Left Ventricular Dysfunction
Keywords: myocardial steatosis; fasting; estrogen; biological sex as a variable
MeSH Terms: conditions — Heart Diseases; Ventricular Dysfunction, Left; Fasting | interventions — Ortho Evra; cetrorelix; Angptl4 protein, mouse; Lower Body Negative Pressure

STUDY DESIGN:
Intervention Model Description: Subjects are studied (bloods and MRI) before and after intervention (2 day fast or 2 day fast with GnRH antagonist and estrogen add back).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Fasting only (Experimental): To acutely elevate myocardial triglyceride content, subjects will be asked to abstain from eating for 2 days (reproducibly causes a significant and physiological increase in myocardial fat deposition, transiently). Subjects will be allowed water and/or an isotonic saline solution in order to maintain hydration status.
  Interventions: Other: Fasting
- LBNP Only (Experimental): Subjects undergo lower body negative pressure at 40 mmHg.
  Interventions: Other: Lower Body Negative Pressure
- Estrogen add back with GnRHant (Experimental): Subjects are given estradiol patch.
  Interventions: Drug: Estradiol patch; Drug: Cetrotide; Other: Fasting
- Placebo add back with GnRHant (Experimental): Subjects are given placebo patch.
  Interventions: Drug: Cetrotide; Other: Fasting

INTERVENTIONS:
Drug: Estradiol patch — Brand name Climara for estrogen add back portion of study. Premenopausal women treated with a GnRH antagonist will be randomized to estrogen add-back or placebo. Thus, for women without contradictions to estrogen use, the risks associated with their use for the duration proposed in these studies (i.e., 6 days) are small. The respective estradiol regimen is a standard approved dose for treatment of hot flashes and the prevention of osteoporosis, and this dose will increase E2 to concentrations typically observed during the mid to late follicular phase of the menstrual cycle.
  Arms: Estrogen add back with GnRHant
Drug: Cetrotide — Premenopausal women will be treated with the gonadotropin-releasing hormone (GnRH) antagonist Cetrorelix for 6 days in order to suppress ovarian sex hormones. Cetrorelix may cause an anaphylactic reaction in volunteers with hypersensitivity to cetrorelix, GnRH or any other GnRH analogs, or extrinsic peptide hormones or mannitol. It may also cause hot flashes, headaches, and nausea. These are typically transient and of mild intensity. These effects are all reversible upon cessation of cetrorelix. Absence of pregnancy will be confirmed before drug administration.
  Arms: Estrogen add back with GnRHant; Placebo add back with GnRHant
Other: Fasting — Subjects will abstain from food for 48 hours. Subjects will be allowed water and/or an isotonic saline solution in order to maintain hydration status.
  Arms: Estrogen add back with GnRHant; Fasting only; Placebo add back with GnRHant
Other: Lower Body Negative Pressure — This test simulates Earth's gravity. The subject will rest on his/her back, with their lower body sealed in an air-tight chamber from the waist down. The chamber is connected to a vacuum that sucks air from the chamber and creates negative pressure inside and around the subject's lower body. As a result, the subject's blood pool shifts towards their legs, away from their chest and arms.
  Other Names: LBNP
  Arms: LBNP Only

SUMMARY:
To test the specific research questions, healthy men and age-matched healthy premenopausal females will be enrolled. Subjects will undergo cardiac magnetic resonance imaging and spectroscopy (MRI/MRS) to evaluate cardiac morphology/function and fat metabolism. To acutely elevate myocardial triglyceride content, subjects will be asked to abstain from eating for 2 days (reproducibly causes a significant and physiological increase in myocardial fat deposition, transiently). Subjects will be allowed water and/or an isotonic saline solution in order to maintain hydration status. After screening, subjects will meet with the research coordinator or an investigator for a discussion, with opportunity for questions, before applicable consent forms are obtained. The subject will be screened for metal in or on their body and claustrophobia using a standard MR screening form. A venous blood sample will be taken for measurement of metabolic health, circulating hormones, and systemic inflammation. Imaging will include cine imaging for global morphology and function, tissue tagging for regional tissue deformation, spectroscopy for fat quantification. After baseline images of the heart are obtained, the subject will be asked to squeeze a MR-safe handgrip dynamometer at 30% of their maximum while images of the heart are obtained. Blood pressure will also be measured at rest and during stress. Each MRI will take approximately 90-120 minutes.

Aim 1 will test the hypothesis that cardiac steatosis induced left ventricular dysfunction is sexually dimorphic, by comparing age-matched men and premenopausal women before and after 48 of fasting. Subjects will complete the MRI/MRS protocol described above before and after the fasting intervention.

Aim 2 will test the hypothesis that estrogen is protective against cardiac steatosis-induced dysfunction, by suppressing ovarian sex hormones with a GnRH antagonist and repeating the fasting studies with and without estrogen add-back. 30 female subjects will be treated with GnRH antagonist and repeat the 48 hour fasting intervention and cardiac MRI/MRS protocol. 15 of the subjects will receive estrogen add-back using a transdermal patch, the other 15 subjects will receive a placebo patch.

Aim 3 will test whether plasma and myocardial fatty acid composition is sexually dimorphic, by performing comprehensive plasma and myocardial lipidomics assessment.

ELIGIBILITY:
Inclusion Criteria:

* blood pressure <140/90 mmHg
* BMI between 18.5 and 30 kg/m2
* sedentary or recreationally active (<3 days of vigorous aerobic exercise each week)
* no use of oral contraceptives hormone therapy, or other medications that might influence cardiovascular function
* nonsmokers.

Exclusion Criteria:

* Women will be excluded with

  1. history of or active estrogen-dependent neoplasms, acute liver or gallbladder disease, vaginal bleeding, venous thromboembolism, hypertriglyceridemia, and CVD
  2. known allergy to transdermal patch, GnRHant (i.e., hypersensitivity to cetrorelix, extrinsic peptide hormones, mannitol, GnRH, benzyl alcohol - the vehicle for injection of cetrorelix)
  3. history of stomach ulcer or bleeding
  4. other contraindications to hormone replacement therapy or GnRHant, (i.e., taking Levodopa, medications that can inhibit folate metabolism including methotrexate).

Other conditions for which individuals will be excluded from the study include:

diabetes active infection history of seizures or disease that affects the nervous system sepsis an abnormal resting ECG contraindications to MRI pregnant or planning to become pregnant smoking history illicit drug use (excluding occasional marijuana).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-09-13 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular relaxation rate | 1 week
  Measured at each of the 4 MRIs by tissue tagging
Comprehensive plasma lipidomics | 1 week
  Measured from blood drawn at each of the 4 MRIs

CONTACTS AND LOCATIONS:
Overall Officials: michael nelson, PhD, Principal Investigator — University of Texas at Arlington
Locations (1):
- University of Texas at Arlington, Arlington, Texas, United States